CLINICAL TRIAL: NCT04746534
Title: Cohort SURVI : Intestinal Ischemia and Vascular Diseases
Acronym: Survibase
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200184
Record Dates: First submitted 2020-12-18; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2020-11

CONDITIONS: Mesenteric Ischemia
MeSH Terms: conditions — Mesenteric Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The first Intestinal Vascular Emergency Unit (SURVI), with the institutional support of AP-HP, opened on 4 January 2016, within the Paris-Nord Val de Seine University Hospital Group. This intensive care is dedicated to the management of mesenteric ischemias (acute mesenteric ischemias, chronic mesenteric ischemias) and Intestinal Vascular Diseases Without Ischemia. The organisation of this type of dedicated centre, combining advances in resuscitation, interventional radiology and knowledge of intestinal vascular diseases, has led to a radical change in the prognosis for acute mesenteric ischaemia with a survival rate of over 80% and an intestinal resection rate of less than 40%.

Acute mesenteric ischaemia (AMI) is characterised by the combination of digestive distress and vascular insufficiency: occlusive (thrombosis, embolism, arterial, venous) or non-occlusive (low flow or vasospasm). The vital prognosis is catastrophic in the absence of treatment (the mortality rate of an intestinal infarction is almost 100% without treatment), and the functional and anatomical after-effects are major for the survivors.

Many intestinal vascular diseases have been identified as providing acute and chronic mesenteric ischaemia. The nosological framework of these diseases is broad, ranging from constitutional diseases of the vessels (collagenosis, arcuate ligament syndrome) to acquired diseases of a thrombophilic, cardiac, degenerative, autoimmune, iatrogenic, traumatic nature... The rarity of these diseases (with the exception of atherosclerotic disease, the incidence of which is increasing with the ageing of the population) makes their level of knowledge insufficient.

The natural history of vascular diseases without ischaemia (rate of acute and chronic mesenteric ischaemia, mortality rate, resection rate...) is currently not described.

The construction of a longitudinal observational cohort is necessary for the prevalence of ischaemic complications and predictive factors.

DETAILED DESCRIPTION:
The first Intestinal Vascular Emergency Unit (SURVI), with the institutional support of AP-HP, opened on 4 January 2016, within the Paris-Nord Val de Seine University Hospital Group. This intensive care is dedicated to the management of mesenteric ischemias (acute mesenteric ischemias, chronic mesenteric ischemias) and Intestinal Vascular Diseases Without Ischemia. The organisation of this type of dedicated centre, combining advances in resuscitation, interventional radiology and knowledge of intestinal vascular diseases, has led to a radical change in the prognosis for acute mesenteric ischaemia with a survival rate of over 80% and an intestinal resection rate of less than 40%.

Acute mesenteric ischaemia (AMI) is characterised by the combination of digestive distress and vascular insufficiency: occlusive (thrombosis, embolism, arterial, venous) or non-occlusive (low flow or vasospasm). The vital prognosis is catastrophic in the absence of treatment (the mortality rate of an intestinal infarction is almost 100% without treatment), and the functional and anatomical after-effects are major for the survivors.

Many intestinal vascular diseases have been identified as providing acute and chronic mesenteric ischaemia. The nosological framework of these diseases is broad, ranging from constitutional diseases of the vessels (collagenosis, arcuate ligament syndrome) to acquired diseases of a thrombophilic, cardiac, degenerative, autoimmune, iatrogenic, traumatic nature... The rarity of these diseases (with the exception of atherosclerotic disease, the incidence of which is increasing with the ageing of the population) makes their level of knowledge insufficient.

The natural history of vascular diseases without ischaemia (rate of acute and chronic mesenteric ischaemia, mortality rate, resection rate...) is currently not described.

The construction of a longitudinal observational cohort is necessary for the prevalence of ischaemic complications and predictive factors.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* IMVI including :
* acute mesenteric ischaemia defined by acute digestive distress in relation to arterial and/or venous, occlusive and/or non-occlusive splanchnic-mesenteric vascular insufficiency, in the absence of an alternative diagnosis

  * Chronic mesenteric ischaemia defined by chronic digestive distress (duration of symptom evolution >30 days) related to occlusive or non- occlusive arterial or venous vascular insufficiency.
  * MVI: gastrointestinal arterial or venous diseases without ischaemia (atheroma, embolism, thrombosis, dissection, mediolysis, aneurysm, dysplasia, sheathing, compression, torsion)

Exclusion Criteria:

* Left ischaemic colitis without damage to the celiac trunk and/or superior mesenteric artery
* Dissection of the abdominal aorta without intestinal ischaemia
* Portal thrombosis without extension to the superior mesenteric vein
* Portal thrombosis without extension to the superior mesenteric vein
* Traumatic rupture of the digestive arteries
* Non-injected abdominal scanner or no abdominal scanner
* Patient opposition to participation in research
* Patient under guardianship / curators
* Vulnerable patient: pregnant or breastfeeding women, persons deprived of their liberty, minors, adults unable or unwilling to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: active patient file of the SURVI service
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2020-11-27 (Actual); Primary Completion 2041-01-04 (Estimated); Study Completion 2041-01-04 (Estimated)

PRIMARY OUTCOMES:
mortality of Intestinal Ischemia | 1 year
  To study the prognosis of Intestinal (acute and chronic) Ischemia and Vascular Diseases (IIVD) at 1 year in terms of mortality.
mortality of Intestinal Ischemia | 5 years
  To study the prognosis of Intestinal (acute and chronic) Ischemia and Vascular Diseases (IIVD) at 5 years in terms of mortality.
Vascular Diseases (IIVD) | 1 year
  To study the prognosis of Intestinal (acute and chronic) Ischemia and Vascular Diseases
Vascular Diseases (IIVD) | 5 years
  To study the prognosis of Intestinal (acute and chronic) Ischemia and Vascular Diseases

SECONDARY OUTCOMES:
Describe the prevalence of IIVD | 1 year
Describe the prevalence of IIVD | 5 years
Study mortality and its associated factors of IIVD | 1 year
Study mortality and its associated factors of IIVD | 5 years
Study the risk of intestinal resection of IIVD and its associated factors. Among resected patients, describe the incidence of short intestinal syndrome and dependence on parenteral nutrition | 1 year
Study the risk of intestinal resection of IIVD and its associated factors. Among resected patients, describe the incidence of short intestinal syndrome and dependence on parenteral nutrition | 5 years
To study the risk of vascular restenosis in all revascularised patients with IIVD and its associated factors | 1 year
To study the risk of vascular restenosis in all revascularised patients with IIVD and its associated factors | 5 years
To study the incidence of recurrence or ischaemic complications (acute or chronic) in IIVD and their associated factors. | 1 year
To study the incidence of recurrence or ischaemic complications (acute or chronic) in IIVD and their associated factors. | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Olivier CORCOS, Clichy, France

IPD SHARING:
Plan to Share IPD: Yes